CLINICAL TRIAL: NCT04320953
Title: Non-contact Endoscopy at Covid-19 Outbreak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ncMCE1
Record Dates: First submitted 2020-03-21; First posted 2020-03-25 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Gastrointestinal Disease; Infectious Disease
MeSH Terms: conditions — Gastrointestinal Diseases; Communicable Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-contact MCE examination (Experimental): Study subject in this arm receives non-contact MCE examination.
  Interventions: Device: Non-contact MCE system

INTERVENTIONS:
Device: Non-contact MCE system — After an overnight fasting and drinking 1000 mL water and simethicone for gastric dilatation and preparation, the study subject positions himself (herself) on the examination bed in Room A, while the operating doctor sits in Room B at the remote control workstation instructing her to swallow the capsule via the audio-visual exchange system. After the capsule entering the stomach, the doctor manipulated the two joysticks on the remote control workstation, mobilizing the robotic magnetic arm, and simultaneously driving the precise movement and rotation of the capsule to perform the gastric examination.

SUMMARY:
The COVID-19 outbreak and spread throughout the world now constitutes a global public health emergency. Direct contact between doctors and patients in daily practice bears potential risk of Covid-19 infection, and telemedicine, or non-contact medicine, in this circumstance, offers an ideal solution. Remote controlling capsule endoscopy system for gastric examination was recently developed and applicated in clinical practice.

DETAILED DESCRIPTION:
The novel non-contact magnetically-controlled capsule endoscopy (MCE) system (Ankon Technologies, China) adds a remote control workstation and a audio-visual exchange system to the original well-establish MCE system, which consists of a robotic magnetic arm, a workstation (now bypassed) and a capsule endoscope, and boasts a 90% sensitivity and 94% specificity for diagnosing gastric focal lesions. This feasibility study aims to evaluate the technical success, clinical success and adverse events of the first clinical application of non-contact MCE system.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consents before joining this study

Exclusion Criteria:

* Dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy
* Refused abdominal surgery to take out the capsule in case of capsule retention
* Implanted pacemaker, except the pacemaker is compatible with MRI
* Other implanted electromedical devices or magnetic metal foreign bodies
* Pregnancy or suspected pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Technical success | During the procedure
  Maneuvarability of the remote control MCE system

SECONDARY OUTCOMES:
Clinical success | During the procedure
  Complete observation of the mucosa (>90% of the mucosa observed) in gastric cardia, fundus, body, angulus, antrum and pylorus
Adverse events | During and within 2 weeks after the procedure
  Adverse events during and after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

REFERENCES:
- [Background] Hollander JE, Carr BG. Virtually Perfect? Telemedicine for Covid-19. N Engl J Med. 2020 Apr 30;382(18):1679-1681. doi: 10.1056/NEJMp2003539. Epub 2020 Mar 11. No abstract available. PMID 32160451
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Zhao AJ, Qian YY, Sun H, Hou X, Pan J, Liu X, Zhou W, Chen YZ, Jiang X, Li ZS, Liao Z. Screening for gastric cancer with magnetically controlled capsule gastroscopy in asymptomatic individuals. Gastrointest Endosc. 2018 Sep;88(3):466-474.e1. doi: 10.1016/j.gie.2018.05.003. Epub 2018 May 9. PMID 29753039
- [Background] Tai FWD, Ching HL, Hale MF, McAlindon ME. Upper gastrointestinal endoscopy: can we cut the cord? Lancet Gastroenterol Hepatol. 2019 Oct;4(10):749-751. doi: 10.1016/S2468-1253(19)30262-6. No abstract available. PMID 31511198
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825